CLINICAL TRIAL: NCT00276133
Title: Effects of Atorvastatin Versus Probucol on Low-Density Lipoprotein Subtype Distribution and Renal Function in Hyperlipidemic Patients With Non-Diabetic Nephropathy
Brief Title: Effects of Atorvastatin Versus Probucol on Small Dense LDL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yokohama City University Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 7332-1
Record Dates: First submitted 2006-01-11; First posted 2006-01-12 (Estimated); Last update posted 2007-05-09 (Estimated); Status verified 2007-05

CONDITIONS: Chronic Nephropathy
Keywords: small dense LDL

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Effects of atorvastatin versus probucol on small dense LDL

SUMMARY:
Small dense low-density lipoprotein (LDL) plays an important role in causing glomerular injury through conversion to an oxidatively modified form of LDL. However, few studies evaluated the effects of antilipidemic agents on the LDL particle size and renoprotective actions in hyperlipidemic patients with non-diabetic nephropathy.

DETAILED DESCRIPTION:
The study is a randomized crossover trial comparing the effect of atorvastatin (10 mg/day) and probucol (500 mg/day) for 24 weeks in 30 patients (urinary albumin excretion 0.3-2.0 g/day, and creatinine clearance > 30 ml/min/1.73 m2 or serum creatinine concentration < 2 mg/L). Lipid parameters, mean LDL particle diameter, creatinine clearance, and urinary albumin to creatinine excretion ratio are measured before and during treatment periods. It will be evaluated that, first, whether atorvastatin and probucol significantly reduce serum total cholesterol and LDL cholesterol concentrations, second, whether atorvastatin and probucol significantly increase the LDL particle size, third, whether significant differences in urinary albumin/creatinine excretion ratio and creatinine clearance are observed in both groups during treatment.

ELIGIBILITY:
Inclusion Criteria:

* Hyperlipidemic patients with non-diabetic nephropathy

Exclusion Criteria:

* Endocrinological, hematological or hepatic disease
* Cerebral infarction or hemorrhage
* Homozygous familial hypercholesterolemia
* Uncontrolled hypertension
* Myocardial infarction occurring within the previous 6 months
* Unstable angina
* Diabetic nephropathy
* Abnormal thyroid function
* Receiving steroids or immunosuppressive agents

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2004-01; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Normalization of serum cholesterol concentrations | One year

CONTACTS AND LOCATIONS:
Overall Officials: Gen Yasuda, MD, Principal Investigator — Yokohama City University Center Hospital
Locations (1):
- Yokohama City University Center Hospital, Yokohama, Kanagawa, Japan

REFERENCES:
- [Background] Yasuda G, Kuji T, Hasegawa K, Ogawa N, Shimura G, Ando D, Umemura S. Safety and efficacy of fluvastatin in hyperlipidemic patients with chronic renal disease. Ren Fail. 2004 Jul;26(4):411-8. doi: 10.1081/jdi-120039826. PMID 15462110